CLINICAL TRIAL: NCT00000386
Title: Behavior Therapy for Childhood OCD
Brief Title: Behavior Therapy for Children and Adolescents With Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01MH058459 (NIH); DSIR CT-S
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Adolescence; Child; Comparative Study; Family; Female; Human; Male; Obsessive-Compulsive Disorder; Relaxation Techniques; Obsessive-Compulsive Disorder -- *therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Relaxation Therapy; Behavior Therapy; Family Therapy

INTERVENTIONS:
Behavioral: Exposure and Response Prevention
Behavioral: Family Treatment Program
Behavioral: Relaxation Training
Behavioral: Behavior therapy
Behavioral: Family Counseling

SUMMARY:
The purpose of this study is to evaluate a behavioral treatment program for children and adolescents with OCD and their families. Exposure and Response Prevention (ERP) behavior therapy, in which the patient is gradually exposed to the object or situation that causes anxiety and is taught to refrain from responding in a compulsive manner, is combined with family counseling (Family Treatment Program). This treatment will be compared to Relaxation Training (RT).

OCD is a long-term, often disabling disorder that can cause significant family disruption. ERP is a promising treatment for children with OCD, and it is thought that family participation (through the Family Treatment Program) may be a helpful addition. RT is a common treatment for anxiety.

Patients are assigned randomly (like tossing a coin) to receive either the ERP/Family Treatment Program or RT. Both treatments will be delivered over 12 90-minute outpatient sessions to youngsters and their families. All participants (patients and family members) will be assessed for treatment response each month during treatment, after treatment is finished, and then at 2 follow-up visits over the following 6 months.

A child/adolescent may be eligible for this study if he/she:

Has obsessive-compulsive disorder (OCD), is medication-free, and is 8 to 17 years old.

DETAILED DESCRIPTION:
To evaluate a standardized multicomponent cognitive behavioral treatment program for child and adolescent obsessive-compulsive disorder (OCD). The treatment program consists of individual Exposure and Response Prevention (ERP) for the OCD child plus a concurrent family intervention designed to reduce OCD-related family conflict, facilitate family disengagement from the affected child's OCD behavior, and rebuild normal family interaction patterns. The ERP/Family Treatment Program is compared with Relaxation Training (RT).

OCD is a chronic, often disabling disorder in childhood that has been associated with increased rates of parental psychopathology and significant disruptions in family relationships and functioning. Preliminary studies suggest that ERP is an effective treatment for children with OCD although no controlled trials to this effect have been published. RT was selected as the comparison treatment because of its credibility as an anxiety treatment and familiarity to potential subjects. RT has been used as a comparison condition for at least 2 randomized controlled ERP trials for adult OCD and shown to be ineffective in treating this disorder. Although it has long been hypothesized that family participation in treatment may be helpful, this is the first controlled study incorporating a systematic manualized family treatment component.

Participants are randomly assigned to receive either the combined ERP/Family Treatment Program (n=56) or RT (n=24). Both treatments are delivered over 12 90-minute outpatient sessions according to detailed treatment manuals.Youth and families undergo comprehensive and systematic, including behavioral, assessments by blind clinical evaluators at baseline, monthly during treatment, post-treatment and 2 follow-up evaluations over 6 months. Treatment outcome is examined in multimodal fashion and across multiple functional domains with a special emphasis on family contextual variables. The impact of baseline functioning, including family context, and initial change over time on treatment outcome is also systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Obsessive-compulsive disorder for which he/she has not received medication.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-12; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Overall Officials: John C. Piacentini, PhD, Principal Investigator
Locations (1):
- Univ. of California / Los Angeles / Neuropsychiatric Inst., Los Angeles, California, United States

REFERENCES:
- [Derived] Kircanski K, Wu M, Piacentini J. Reduction of subjective distress in CBT for childhood OCD: nature of change, predictors, and relation to treatment outcome. J Anxiety Disord. 2014 Mar;28(2):125-32. doi: 10.1016/j.janxdis.2013.05.004. Epub 2013 May 21. PMID 23774008
- [Derived] Piacentini J, Bergman RL, Chang S, Langley A, Peris T, Wood JJ, McCracken J. Controlled comparison of family cognitive behavioral therapy and psychoeducation/relaxation training for child obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1149-61. doi: 10.1016/j.jaac.2011.08.003. Epub 2011 Sep 22. PMID 22024003